CLINICAL TRIAL: NCT03468686
Title: The Study of Effectiveness of Unilateral and Bilateral Repetitive Transcranial Magnetic Stimulation (rTMS) on Rumination and Anhedonia in Patients With Major Depressive Disorder
Brief Title: The Study of Effectiveness of rTMS on Rumination and Anhedonia in Patients With Major Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tehran (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, reza kazemi, Researcher, University of Tehran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4748
Record Dates: First submitted 2018-02-06; First posted 2018-03-16 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Major Depressive Disorder; Bipolar Depression
Keywords: MDD; rTMS; Rumination; Anhedonia
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder; Rumination Syndrome; Anhedonia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- bilateral rTMS (Active Comparator): sequential bilateral repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Bilateral rTMS
- Sham rTMS (Sham Comparator): Sham Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Sham rTMS
- Unilateral rTMS (Active Comparator): Unilateral (High frequency) repetitive Transcranial Magnetic Stimulation (rTMS)
  Interventions: Device: Unilateral rTMS (High frequency)

INTERVENTIONS:
Device: Bilateral rTMS — The coil will locate on F3 and F4 in accordance with the 10-20 international system. bilateral rTMS include stimulate the right DLPFC at 1 Hz for a 10 seconds train of stimulation, and a total of 150 pulse trains. Immediately after that, the stimulation was carried out on the left DLPFC at 10 Hz, 5 seconds of stimulation, with 10 second inter-train interval and 75 pulse trains.
  Arms: bilateral rTMS
Device: Sham rTMS — The same parameters will use in the sham rTMS. However, the coil adjust at an angle of 90º vertically on the skull in a way that one wing place on the head.
  Arms: Sham rTMS
Device: Unilateral rTMS (High frequency) — The coil will locate on F3 in accordance with the 10-20 international system. Unilateral rTMS include stimulate the Left DLPFC at 10Hz for a 5seconds train of stimulation, 10 seconds inter-train interval, and a total of 75 pulse trains. .
  Arms: Unilateral rTMS

SUMMARY:
Rumination is significantly frequent in major depressive disorder. However, not a lot of studies have investigated the effects of repetitive transcranial magnetic stimulation on rumination and its electrophysiological correlates. This study recruited 61 participants who were randomly assigned to sham, bilateral, or unilateral stimulation groups to investigate the potential differences between these stimulation protocols and changes in the behavioral and electrophysiological outcomes after treatment.

DETAILED DESCRIPTION:
This study aims to compare the effect of unilateral and bilateral rTMS on the reduction of rumination and anhedonia and their associated neural networks. In a randomized double-blind trial, 65 patients with depressive disorder in Atieh Clinical Neuroscience Center are assigned to three groups. The first group receives bilateral rTMS for 20 sessions on right and left DLPFC; the second group receives unilateral rTMS for 20 sessions on LDLPFC; third group receives sham rTMS for 10 sessions. In this group, the stimulation parameters are similar to that in the actual rTMS group, except that the coil angel is 90° and perpendicular to the head. Rumination and anhedonia symptoms will be measured by the Ruminative Responses Scale (RRS) and Snaith-Hamilton Pleasure Scale (SHAPS) in the baseline and after the 20th session. In order to investigate the neural networks associated with rumination and anhedonia, EEG of patients will be recorded at the first session and at the end of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients male and female with the range of 18-65 years of age
* The diagnosis of Major depressive disorder according to DSM-V
* Having BDI>18
* Having stable symptoms as defined by not requiring a change in medication for at least 4 weeks
* Completion of consent form
* Being under supervision of a psychiatrist

Exclusion Criteria:

* The history of rTMS treatment for any reason
* Cardiac pacemaker
* The risk of seizure with any reasons
* Pregnancy
* High risk of suicide
* Intracranial implant and other ferromagnetic materials close to the head

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2016-12-21 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Rumination Symptoms | baseline before start of treatment and immediately after the last treatment session.
  The Ruminative Responses Scale (RRS) is a measure of depressive rumination which has two subscales: Both subscales are composed of five items. Brooding and Reflection. Higher score indicate a higher level of ruminative responses (range: 22-88).
changes in default mode network | baseline before start of treatment and immediately after the last treatment session.
  EEG
Anhedonia Symptoms | baseline before start of treatment and immediately after the last treatment session.
  Snaith-Hamilton Pleasure Scale (SHAPS), a measure of anhedonia

SECONDARY OUTCOMES:
Depressive symptoms measured by the 17-item Hamilton Depression Rating Scale | baseline before start of treatment and immediately after the last treatment session.
  Hamilton Depression Rating Scale (HDRS),(HRSD17) Range: 0-53 Normal: 0-7 Mild: 8 - 13 Moderate 14 - 18 Severe: 19-22 Very severe > 22
Depressive symptoms measured by the 21-item Beck Depression Inventory-II | baseline before start of treatment and immediately after the last treatment session.
  Beck Depression Inventory-II (BDI-II), (BDI-II) Range: 0-63 Normal: 0-13 Mild: 14- 9 Moderate 20- 28 Severe: 29-63

CONTACTS AND LOCATIONS:
Overall Officials: Reza Kazemi, PhD, Principal Investigator — Atieh Clinical Neuroscience center
Locations (1):
- Atieh Clinical Neuroscience Center (ACNC), Tehran, Iran

REFERENCES:
- [Result] Kazemi R, Rostami R, Nasiri Z, Hadipour AL, Kiaee N, Coetzee JP, Philips A, Brown R, Seenivasan S, Adamson MM. Electrophysiological and behavioral effects of unilateral and bilateral rTMS; A randomized clinical trial on rumination and depression. J Affect Disord. 2022 Nov 15;317:360-372. doi: 10.1016/j.jad.2022.08.098. Epub 2022 Aug 30. PMID 36055535